CLINICAL TRIAL: NCT04116905
Title: Intensive Lifestyle Interventions for Remission of Metabolic Syndrome in Overweight or Obese Individuals
Brief Title: Intensive Lifestyle Intervention for Remission of Metabolic Syndrome
Acronym: INSLIMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIMS
Record Dates: First submitted 2019-09-16; First posted 2019-10-07 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2019-09

CONDITIONS: Metabolic Syndrome
Keywords: Metablolic syndrome; remission; life style; weight loss
MeSH Terms: conditions — Metabolic Syndrome; Weight Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Lifestyle Intervention (Experimental): Participants randomized to the intensive lifestyle intervention arm will receive a structured, multi-component program consisting of both individualized counseling and group-based sessions. This intervention is specifically designed to facilitate achievement of a clinically significant 15% weight reduction and support long-term weight maintenance."
  Interventions: Behavioral: Intensive Lifestyle Intervention
- Conventional Treatment (Active Comparator): Participants in the conventional treatment arm receive structured group-based education sessions focusing on metabolic syndrome management principles and peer support, with the therapeutic goal of achieving a modest 7% weight reduction
  Interventions: Behavioral: Conventional Treatment

INTERVENTIONS:
Behavioral: Intensive Lifestyle Intervention — The intensive lifestyle intervention program employs a structured, multi-component approach under professional supervision to achieve and sustain 15% weight reduction from baseline. This 12-month intervention features:
  1. A weight loss phase (months 1-5) incorporating: Individualized calorie restriction using partial meal replacement (carbohydrate energy supply ratio is 20~25%, and the daily calorie intake is 22.5*70% kcal/kg/d); exercise recommends at least 150 min of moderate intensity and 2 to 3 resistance training per week; with monthly follow-ups.
  2. A maintenance phase (months 6-12) focusing on: A Healthy, balanced diet, total daily calorie intake is 20-25 kcal/kg/d; exercise recommendations at least 150 minutes of moderate intensity and 2-3 resistance training per week; with follow-ups every 2 months.
  3. Digital health integration: Mobile application-based monitoring of metabolic parameters; real-time feedback and adherence tracking.
  Arms: Intensive Lifestyle Intervention
Behavioral: Conventional Treatment — The conventional treatment arm receive standardized metabolic syndrome management through monthly group education sessions and peer support, with a target of 7% weight reduction from baseline. The program incorporates:
  1. A weight loss phase (months 1-5) incorporating:
     Structured lifestyle education; limit the total energy diet (total daily calorie intake is 22.5*85% kcal/kg/d), with carbohydrates, fat, proteins accounting for 45-55%, 20-30%, and 20-30%, respectively, for the daily energy intake.; physical activity(150 min medium intensity exercise and 2 to 3 resistance training); with monthly follow-ups;
  2. A maintenance phase (months 6-12) focusing on:
     Healthy balanced diet, total daily calorie intake is 20~25 kcal/kg/d; physical activity(150 min medium intensity exercise and 2 to 3 resistance training);with follow-ups every 2 months;
  3. Digital health integration:
  Mobile application-based monitoring of metabolic parameters; real-time feedback and adherence tracking.
  Arms: Conventional Treatment

SUMMARY:
This is a randomized, prospective clinical trial investigating metabolic syndrome in overweight or obese Chinese individuals. The study aims to evaluate the efficacy of a structured intensive lifestyle intervention program in achieving significant weight reduction (targeting 15% weight loss) and promoting metabolic syndrome remission. Additionally, the research will explore the potential mechanisms underlying these therapeutic effects. Furthermore, this study enables phased presentation of the findings.

DETAILED DESCRIPTION:
Background:

Metabolic syndrome is a global public health concern, with prevalence rates ranging from 10% to 84% across different populations. It is strongly associated with multiple chronic non-communicable diseases, including type 2 diabetes, cardiovascular diseases, non-alcoholic fatty liver disease, polycystic ovary syndrome, and certain cancers. Notably, obesity plays a central role in the development of metabolic syndrome, and substantial evidence supports the benefits of significant weight loss in improving its components. Currently, there is a lack of research on lifestyle interventions aimed at weight loss to alleviate metabolic syndrome in affected populations.

Study Design:

This study is a single-center, prospective, randomized controlled trial. Metabolic syndrome (MetS) subjects aged 18-60 years were enrolled and randomly assigned to either an intensive lifestyle intervention group (a low-carbohydrate diet combined with physical exercise, target weight loss of 15%) or a conventional lifestyle intervention group ( energy-restricted diet combined with physical exercise, target weight loss of 7%). Participants underwent a 5-month weight-loss intervention (with monthly follow-ups) followed by a 7-month weight-maintenance phase (with follow-ups every 2 months). During the follow-up period, anthropometric and laboratory parameters were regularly monitored.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 27-45 kg/m2
* Metabolic syndrome: meet at least 3 of the following 5 criteria: waist circumference ≥85 cm (male) or 80 cm (female); TG ≥1.7 mmol/L or with lipid-lowering treatment; HDL<1.04 mmol/L(male) /1.3 mmol/L (female)；SBP ≥ 130 mmHg and / or DBP ≥ 85 mmHg and / or with diagnosed hypertension and anti-hypertensive treatment; fasting glucose ≥ 5.6 mmol/L and / or with diagnosed type 2 diabetes and hypoglycemic treatment. (If with type 2 diabetes, the process of the disease should not exceed 6 years, with the level of C-P ≥3/4 of the lower limit of limit; if with hypertension, BP ≤ 180/110 mmHg without anti-hypertensive agent, or BP ≤160/100 mmHg with 1-2 kinds of anti-hypertensive agents, or BP ≤140/90 mmHg with 3-4 kinds of anti-hypertensive agents; if with hyper-triglyceridemia, TG ≤ 11.2 mmol/L without lipid-lowering agent, or TG ≤ 5.6 mmol/L with lipid-lowering agent.)
* Han Chinese
* Willingness to participate

Exclusion Criteria:

* Participants with metabolic syndrome caused by other secondary factors (genetic diseases related to obesity and hyperlipidemia, Cushing's syndrome, drug-induced obesity and etc.);
* Participants whose body weight fluctuated by more than 5 kg in the last 6 months; who trying to lose weight in the last 3 months; who had used anti-obesity drugs, oral contraceptive, or glucocorticoids in the last 3 months;
* Participants with Type 1 diabetes or gestational diabetes or other types of diabetes;
* Participants with BP ≥ 180/110 mmHg, or malignant hypertension;
* Participants with previous severe gastrointestinal diseases;
* Participants with significant dysfunction of heart, liver, kidney and systemic organs (NYHA Class III or IV; ALT and / or AST ≥ 4 times the normal upper limit; GFR < 60 ml/min) or with malignant tumor;
* Participants with drug abuse or alcohol addiction; with serious mental and neurological disorders;
* Pregnant or lactating women; those who have planned to give birth within the past 1 year;
* Participants with special dietary requirements, or with soy products, milk and other daily food allergies;
* Participants in other clinical trials.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
The remission rate of metabolic syndrome | 12 months
  Participants are considered to have achieved metabolic syndrome remission when they meet ≤2 of the following 5 diagnostic criteria:
  1. Waist circumference ≥85 cm (men) / ≥80 cm (women);
  2. Fasting triglycerides ≥1.7 mmol/L or current lipid-lowering therapy;
  3. HDL cholesterol <1.04 mmol/L (men) / <1.30 mmol/L (women);
  4. Systolic BP ≥130 mmHg and/or diastolic BP ≥85 mmHg, or diagnosed hypertension with antihypertensive treatment;
  5. Fasting glucose ≥5.6 mmol/L, or diagnosed type 2 diabetes with glucose-lowering treatment.
  Remission is defined as sustained resolution of ≥3 criteria.
The proportion of participants achieving 15% weight loss from baseline | 12 months
  The proportion of participants achieving 15% weight loss from baseline

SECONDARY OUTCOMES:
Remission of hypertension | 12 months
  The proportion of participants achieving target blood pressure control (either <130/85 mmHg or <140/90 mmHg) without antihypertensive medication.
Remission of hyperglycemia | 12 months
  The proportion of participants achieving fasting plasma glucose <5.6 mmol/L without glucose-lowering medication.
Remission of hypertriglyceridemia | 12 months
  The proportion of participants achieving triglyceride levels <1.7 mmol/L without lipid-lowering therapy.
Remission of low HDL-C | 12 months
  The sex-specific proportion achieving therapeutic HDL-C targets (≥1.04 mmol/L in males; ≥1.30 mmol/L in females) without lipid-modifying therapy.
Remission of central obesity | 12 months
  Proportion meeting gender-stratified waist circumference criteria (males <85 cm; females <80 cm).

CONTACTS AND LOCATIONS:
Overall Officials: Pengfei Shan, MD, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Yuezhong Ren, MD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China